CLINICAL TRIAL: NCT03803943
Title: Early Communication Intervention for Toddlers With Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Megan Roberts, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DC016877-01A1 (NIH)
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Bilateral
Keywords: Hearing Loss; Toddlers; Early Intervention; Parent-mediated intervention
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Children will enroll in the study around 12 months of age and will be randomly assigned to either a parent-implemented communication intervention (PICT) or a control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and coders will be naive to experimental condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent-Implemented Communication Intervention (PICT) (Experimental): Participants assigned to the PICT condition will receive weekly hour long intervention sessions in their home for 6 months. Parents will learn four sets of communication support strategies: (a) visual (e.g., modeling language within the child's line of sight), (b) interactive (e.g., following the child's attentional focus), (c) responsive (e.g., responding to all communicative attempts), and (d) linguistically stimulating (e.g., modeling language targets, expanding child communication).
  Interventions: Behavioral: Parent-Implemented Communication Intervention (PICT)
- No Intervention - Business-as-usual control (Placebo Comparator): Participants assigned to the BAU control group will not receive the PICT intervention.
  Interventions: Other: No Intervention - Business-as-usual control

INTERVENTIONS:
Behavioral: Parent-Implemented Communication Intervention (PICT) — Weekly hour long intervention sessions for 6 months
  Other Names: PICT
  Arms: Parent-Implemented Communication Intervention (PICT)
Other: No Intervention - Business-as-usual control — Does not receive PICT intervention
  Other Names: BAU
  Arms: No Intervention - Business-as-usual control

SUMMARY:
Improving spoken language outcomes for children with hearing loss has important public health implications. This is a randomized clinical trial of 96 children with hearing loss that examines the effects of a parent-implemented early communication intervention on prelinguistic and spoken language outcomes. The study is open for national recruitment. Parents participate via video call with their child and receive technology to assist with virtual visits.

DETAILED DESCRIPTION:
While children with hearing loss (HL) are experiencing greater gains in spoken language than ever before, considerable variability exists and many children with HL continue to have poorer language skills than their hearing peers. Critical to reducing this variability is the identification of: (a) effective early communication interventions for children with HL and (b) child and parent characteristics that influence intervention outcomes (moderators and mediators). However, to date, only the pilot study for this proposed study has directly examined the effects of an early communication intervention for children with HL within the context of a randomized clinical trial. The overarching goals of the proposed study are to: (a) evaluate the effects of teaching parents to use communication support strategies on child communication outcomes and (b) examine parent and child characteristics that moderate and mediate intervention outcomes. The central hypothesis is that systematic parent training will result in greater parental use of communication support strategies, greater child pre-symbolic communicative acts, and greater child spoken language outcomes. The specific aims include: (a) comparing parent use of communication support strategies and child pre-symbolic communicative acts between intervention and control groups during and immediately following intervention (from 12 to 18 months of age), (b) examining parent (identification of child communication) and child (sensitivity to social contingency; attention to speech) moderators of intervention outcomes; (c) comparing parent use of communication support strategies and child spoken language outcomes between intervention and control groups after intervention (from 18 and 36 months of age); and (d) examining parent (use of communication support strategies) and child (pre-symbolic communicative acts) mediators of intervention outcomes. The proposed study will enroll 96 children with mild to profound bilateral hearing loss. Children will enroll in the study around 12 months of age and will be randomly assigned to either a parent-implemented communication intervention (PICT) or a control group. Children in both groups will be assessed: (a) at 12 months of age (immediately before intervention), (b) at 18 months of age (immediately after intervention), and (c) at 36 months of age (18 months after the end of intervention). Children in the intervention group will receive weekly, 1-hour intervention sessions for 6-months that: (a) are delivered during an important prelinguistic period of language development, (b) incorporate visual, interactive, responsive, and linguistically stimulating communication support strategies that are associated with stronger language skills in children with HL, and (c) include systematic parent training found to be effective in teaching parents to use communication support skills in children with language delays. The proposed research is significant because effective early communication intervention is likely to reduce persistent language delays in children with HL, thereby advancing the field of childhood hearing loss, where there is a striking paucity of rigorous communication intervention research.

ELIGIBILITY:
Inclusion Criteria:

* have bilateral, congenital HL as measured by a review of medical records
* enrollment in the study between 12 and 18 months of age
* have no known additional disabilities (e.g., Down syndrome, cerebral palsy, seizure disorder, blindness, etc.) as measured by review of medical records and parent report
* have English as the primary language spoken at home
* have one parent with normal hearing, and (f) are exposed to some degree of spoken language by their parents (total communication, auditory/oral)

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Y Roberts, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and associated documentation available to users only under a data-sharing agreement that provides for a commitment: (1) to use the data only for research purposes and not to identify any individual participant; (2) to secure the data using appropriate computer technology; (3) to destroy or return the data after analyses are completed; and (4) to cite the grant and key publications describing the database and measures in any resulting presentations and publications.
Access Criteria: Transcripts from caregiver-child and examiner-child language samples will also be donated to the Child Language Data Exchange System (http://childes.psy.cmu.edu), an international repository of child language data. Access to the data will be openly available. Researchers who access the transcripts will be expected to abide by the established guidelines for use of TalkBank data http://talkbank.org/share/irb/options.html.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization occurred at the dyad level, with each dyad consisting of one parent and one child. The dyad was considered the enrolled unit in the study, and each dyad was randomly assigned to either the intervention or control group. The arm/group title is labeled based on the dyad's assignment and reflects the joint participation of both caregiver and child.
Groups:
- Parent-Implemented Communication Intervention (PICT) - Children; Parent-Implemented Communication Intervention (PICT) - Parents: Participants assigned to the PICT condition will receive weekly hour long intervention sessions in their home for 6 months. Parents will learn four sets of communication support strategies: (a) visual (e.g., modeling language within the child's line of sight), (b) interactive (e.g., following the child's attentional focus), (c) responsive (e.g., responding to all communicative attempts), and (d) linguistically stimulating (e.g., modeling language targets, expanding child communication).
  Parent-Implemented Communication Intervention (PICT): Weekly hour long intervention sessions for 6 months
- No Intervention - Business-as-usual control - Children; No Intervention - Business-as-usual control - Parents: Participants assigned to the BAU control group will not receive the PICT intervention.
  No Intervention - Business-as-usual control: Does not receive PICT intervention
Period: Overall Study
Arm/Group | Parent-Implemented Communication Intervention (PICT) - Children | No Intervention - Business-as-usual control - Children | Parent-Implemented Communication Intervention (PICT) - Parents | No Intervention - Business-as-usual control - Parents
Started | 48 | 46 | 48 | 46
Completed | 46 | 44 | 46 | 44
Not Completed | 2 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: 94 parent-child dyads were randomized at baseline, 46 of whom were allocated to the PICT group and 48 of whom were randomized to the BAU control group.
Groups:
- Parent-Implemented Communication Intervention (PICT): Children; Parent-Implemented Communication Intervention (PICT): Parents: Participants assigned to the PICT condition will receive weekly hour long intervention sessions in their home for 6 months. Parents will learn four sets of communication support strategies: (a) visual (e.g., modeling language within the child's line of sight), (b) interactive (e.g., following the child's attentional focus), (c) responsive (e.g., responding to all communicative attempts), and (d) linguistically stimulating (e.g., modeling language targets, expanding child communication).
  Parent-Implemented Communication Intervention (PICT): Weekly hour long intervention sessions for 6 months
- No Intervention - Business-as-usual control: Children; No Intervention - Business-as-usual control: Parents: Participants assigned to the BAU control group will not receive the PICT intervention.
  No Intervention - Business-as-usual control: Does not receive PICT intervention
- Total: Total of all reporting groups
Arm/Group | Parent-Implemented Communication Intervention (PICT): Children | No Intervention - Business-as-usual control: Children | Parent-Implemented Communication Intervention (PICT): Parents | No Intervention - Business-as-usual control: Parents | Total
Number analyzed (Participants) | 46 | 48 | 46 | 48 | 188
Age, Continuous [Mean (Standard Deviation); unit: months] — Age of the child participant Population: This is a baseline measure of the child participants only.
  months
    number analyzed (Participants) | 46 | 48 | 0 | 0 | 94
    (all) | 15.6 (1.8) | 15.5 (2.1) |  |  | 15.6 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 34 | 43 | 43 | 146
  Male | 20 | 14 | 3 | 5 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 6 | 7 | 28
  Not Hispanic or Latino | 39 | 38 | 40 | 37 | 154
  Unknown or Not Reported | 0 | 2 | 0 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 5 | 3 | 5 | 2 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 4 | 1 | 10
  White | 30 | 39 | 31 | 40 | 140
  More than one race | 6 | 2 | 1 | 1 | 10
  Unknown or Not Reported | 1 | 2 | 5 | 4 | 12
Total Number of Communicative Acts from the Language Sample - Child [Mean (Standard Deviation); unit: Total Weighted Frequency Score] — During the 10-minute interaction, the child played with toys and wordless picture books. A research assistant transcribed and coded all communicative acts. Each communicative act was assigned a weight reflecting its developmental complexity: gestures and vocalizations = 1 point, single words = 2 points, and multiple-word utterances = 3 points. The Total Weighted Frequency Score (Min = 0, Max = NA) is the sum of the weighted frequency of each act, with higher scores reflecting more frequent and complex communicative acts. Population: This is a baseline measure of the child participants only.
  Total Weighted Frequency Score
    number analyzed (Participants) | 46 | 48 | 0 | 0 | 94
    (all) | 54.7 (30.0) | 49.0 (32.6) |  |  | 51.8 (31.3)
Communication and Symbolic Behavior Scales Score - Child [Mean (Standard Deviation); unit: units on a scale] — The child is presented with 6 different activities (wind-up toy, balloon, bubbles, jar, books, play) designed to elicit child communication. The interaction is video recorded and then scored for 20 items across 7 communication scales (emotion and eye gaze, communication, gestures, sounds, words, understanding, and object use). The weighted raw scores for each of the 7 scales were grouped into 3 clusters (social, speech, and symbolic) and combined into a total raw score (min = 0; max = 113). Higher scores indicate better skills. Population: This is a baseline measure of the child participants only.
  units on a scale
    number analyzed (Participants) | 46 | 48 | 0 | 0 | 94
    (all) | 67.5 (24.7) | 58.7 (23.6) |  |  | 63.0 (24.4)
Use of Communication Support Strategies - Parent [Mean (Standard Deviation); unit: units on a scale] — Parent use of communication support strategies was measured from a 12-minute parent-child interaction in which the dyad plays using a standard set of toys. Interactions were video recorded and coded for 13 items representing subcomponents of seven communication support strategies. Each item was rated on a 5-point scale (1 = novice use, 5 = expert use), reflecting the quality and proficiency of parent strategy use. Items were averaged to yield a Total Composite Score (Min = 1, Max = 5), with higher scores indicating more proficient and consistent use of communication strategies. Population: This is a baseline measure of the parent participants only.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 46 | 48 | 94
    (all) |  |  | 3.10 (0.40) | 3.0 (0.40) | 3.10 (.50)
Hearing Level - Child [Count of Participants; unit: Participants] — Hearing level of child participant Population: This is a baseline measure of the child participants only.
  Participants
    number analyzed (Participants) | 46 | 48 | 0 | 0 | 94
    slight | 1 | 2 |  |  | 3
    mild | 9 | 9 |  |  | 18
    moderate | 3 | 9 |  |  | 12
    moderately severe | 11 | 5 |  |  | 16
    severe | 7 | 6 |  |  | 13
    profound | 14 | 17 |  |  | 31
    unknown | 1 | 0 |  |  | 1
Communication Mode - Child [Count of Participants; unit: Participants] — Communication mode of the child participant Population: This is a baseline measure of the child participants only.
  Participants
    number analyzed (Participants) | 46 | 48 | 0 | 0 | 94
    Sign | 14 | 17 |  |  | 31
    No Sign | 32 | 31 |  |  | 63
Hearing Device - Child [Count of Participants; unit: Participants] — Hearing device of the child participant Population: This is a baseline measure of the child participants only.
  Participants
    number analyzed (Participants) | 46 | 48 | 0 | 0 | 94
    Cochlear Implant/Bone Conduction | 24 | 28 |  |  | 52
    Hearing Aid | 22 | 20 |  |  | 42

OUTCOME MEASURES:

1. Primary Outcome: Use of Communication Support Strategies - Parent
Description: Parent use of communication support strategies was measured from a 12-minute parent-child interaction in which the dyad plays using a standard set of toys. Interactions were video recorded and coded for 13 items representing subcomponents of seven communication support strategies. Each item was rated on a 5-point scale (1 = novice use, 5 = expert use), reflecting the quality and proficiency of parent strategy use. Items were averaged to yield a Total Composite Score (Min = 1, Max = 5), with higher scores indicating more proficient and consistent use of communication strategies.
Time Frame: Change from Baseline to Month 7
Population: This is an outcome measure of the parent participants only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent-Implemented Communication Intervention (PICT): Parents | No Intervention - Business-as-usual control: Parents
Number analyzed (Participants) | 46 | 48
units on a scale | .60 (.52) | .02 (.51)

2. Primary Outcome: Total Number of Communicative Acts From the Language Sample - Child
Description: During the 10-minute interaction, the child played with toys and wordless picture books. A research assistant transcribed and coded all communicative acts. Each communicative act was assigned a weight reflecting its developmental complexity: gestures and vocalizations = 1 point, single words = 2 points, and multiple-word utterances = 3 points. The Total Weighted Frequency Score (Min = 0, Max = NA) is the sum of the weighted frequency of each act, with higher scores reflecting more frequent and complex communicative acts.
Time Frame: Change from Baseline to Month 7
Population: This is an outcome measure of the child participants only.
Measure: Mean (Standard Deviation); unit: Total Weighted Frequency Score
Arm/Group | Parent-Implemented Communication Intervention (PICT): Children | No Intervention - Business-as-usual control: Children
Number analyzed (Participants) | 46 | 48
Total Weighted Frequency Score | 57.8 (57.8) | 25.24 (50.1)

3. Primary Outcome: Communication and Symbolic Behavior Scales Score - Child
Description: The child is presented with 6 different activities (wind-up toy, balloon, bubbles, jar, books, play) designed to elicit child communication. The interaction is video recorded and then scored for 20 items across 7 communication scales (emotion and eye gaze, communication, gestures, sounds, words, understanding, and object use). The weighted raw scores for each of the 7 scales were grouped into 3 clusters (social, speech, and symbolic) and combined into a total raw score (min = 0; max = 113). Higher scores indicate better skills.
Time Frame: Month 7
Population: This is an outcome measure of the child participants only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent-Implemented Communication Intervention (PICT): Children | No Intervention - Business-as-usual control: Children
Number analyzed (Participants) | 46 | 48
units on a scale | 104.98 (24.49) | 92.24 (29.61)

4. Secondary Outcome: Use of Communication Support Strategies - Parent
Description: as for outcome 1
Time Frame: Change from Baseline to Month 24
Population: This is an outcome measure of the parent participants only.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Parent-Implemented Communication Intervention (PICT): Parent: Participants assigned to the PICT condition will receive weekly hour long intervention sessions in their home for 6 months. Parents will learn four sets of communication support strategies: (a) visual (e.g., modeling language within the child's line of sight), (b) interactive (e.g., following the child's attentional focus), (c) responsive (e.g., responding to all communicative attempts), and (d) linguistically stimulating (e.g., modeling language targets, expanding child communication).
  Parent-Implemented Communication Intervention (PICT): Weekly hour long intervention sessions for 6 months
- No Intervention - Business-as-usual control: Parent: Participants assigned to the BAU control group will not receive the PICT intervention.
  No Intervention - Business-as-usual control: Does not receive PICT intervention
Arm/Group | Parent-Implemented Communication Intervention (PICT): Parent | No Intervention - Business-as-usual control: Parent
Number analyzed (Participants) | 46 | 48
units on a scale | .30 (.59) | .09 (.58)

5. Secondary Outcome: Spoken Words - Child
Description: Total number of spoken words will be collected using two measures that will be combined used confirmatory factory analysis. Total Number of Words Said from the MacArthur-Bates Communicative Development Inventory: Words and Sentences and the total number of different spoken word roots from a 10-minute language sample in which an assessor plays with the child following a standardized protocol.
Time Frame: Change from Baseline to Month 24
Reporting Status: Not Posted

6. Secondary Outcome: Expressive Communication Standard Score on the Preschool Language Scale - 5th Edition - Child
Description: The child is presented with different receptive tasks, such as following simple directions and pointing to pictures, until the child provides an incorrect response to six consecutive items. A total standard score is calculated based on the raw score and the child's age (min = 50; max = 150). Higher score indicate better outcomes.
Time Frame: Month 24
Population: This is an outcome measure of the child participants only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent-Implemented Communication Intervention (PICT): Children | No Intervention - Business-as-usual control: Children
Number analyzed (Participants) | 46 | 48
units on a scale | 100.44 (20.05) | 93.81 (20.45)

7. Secondary Outcome: Auditory Comprehension Standard Score on the Preschool Language Scale - 5th Edition - Child
Description: The child is presented with different expressive tasks, such as labeling pictures, until the child provides an incorrect response to six consecutive items. A total standard score is calculated based on the raw score and the child's age (min = 50; max = 150). Higher Scores indicate better outcomes.
Time Frame: Month 24
Population: This is an outcome measure of the child participants only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Parent-Implemented Communication Intervention (PICT): Children | No Intervention - Business-as-usual control: Children
Number analyzed (Participants) | 46 | 48
units on a scale | 102.46 (20.27) | 92.14 (23.8)

ADVERSE EVENTS:
Time Frame: Monthly over 18 months
Arm/Group | Parent-Implemented Communication Intervention (PICT): Children | No Intervention - Business-as-usual control: Children | Parent-Implemented Communication Intervention (PICT): Parents | No Intervention - Business-as-usual control: Parents
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48 | 0/46 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48 | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/46 | 1/48 | 0/46 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parent-Implemented Communication Intervention (PICT): Children (N=46) | No Intervention - Business-as-usual control: Children (N=48) | Parent-Implemented Communication Intervention (PICT): Parents (N=46) | No Intervention - Business-as-usual control: Parents (N=48)
Crying (Psychiatric disorders) | 0 (0) | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT03803943/Prot_001.pdf
  • Statistical Analysis Plan (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT03803943/SAP_002.pdf
  • Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03803943/ICF_000.pdf